CLINICAL TRIAL: NCT04227587
Title: Zero-time Exercise on Inactive Adults With Insomnia Disorder: A Randomized Controlled Trial and Mixed-method Process Evaluation
Brief Title: Effects of Zero-Time Exercise (ZTEx) on Inactive Adults With Insomnia Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, YEUNG Wing Fai, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZTXI
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Insomnia, Primary
Keywords: insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zero Time Exercise training (Experimental): Subjects in this group will attend two 2-hour ZTEx training lessons. Each subject will receive a handout and an exercise log. The handout includes a picture-illustrating ZTEx step-by-step protocol. The exercise log is for them to record their time spending on performing the ZTEx.
  Interventions: Other: Zero Time Exercise
- Sleep hygiene education (Active Comparator): Subjects in this group will receive two 2-hour lessons of sleep hygiene education delivered by a registered nurse. Each subject will receive a handout and a sleep hygiene log.Subjects will be told to record their daily compliance with sleep hygiene instructions using yes/no questions in the sleep hygiene log.
  Interventions: Other: Sleep hygiene education

INTERVENTIONS:
Other: Zero Time Exercise — Zero Time Exercise encourage people to increase physical exercise by simple movements that can be done any time at any places. We offer a 2-session training course to train the subjects to do zero-time exercise.
  Arms: Zero Time Exercise training
Other: Sleep hygiene education — We offer a 2-session education course to teach the subjects about sleep hygiene practice.
  Arms: Sleep hygiene education

SUMMARY:
This randomized controlled trial (RCT) with a longitudinal mixed-method process evaluation aims to (1) determine the effectiveness of a ZTEx intervention program, which is a lifestyle-integrated physical activity program, on sleep and related outcomes in inactive adults with insomnia disorder

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) with a longitudinal mixed-method process evaluation aims to (1) determine the effectiveness of a ZTEx intervention program, which is a lifestyle-integrated physical activity program, on sleep and related outcomes in inactive adults with insomnia disorder; (2) identify the facilitators and barriers of ZTEx adherence, (3) explore the possible mechanisms of impact on ZTEx adherence and the same abovementioned outcomes.

This RCT consists of two phases. In the first phase (baseline to week 8), 136 subjects will be randomly allocated to the ZTEx intervention or the sleep hygiene education (SHE) comparison group. They will receive two 2-hour ZTEx training or SHE lessons and practice ZTEx or follow the sleep hygiene instruction for 24 weeks. After assessment at week 8, for the second phase of the study (weeks 9-24), which is a proof-of-concept pilot nested in the RCT, subjects in the ZTEx group will be randomly divided into either an ZTEx with WhatsApp reminder (ZTEx+R) subgroup or an ZTEx without WhatsApp reminder (ZTEx alone) subgroup to evaluate the effects of WhatsApp reminders on exercise adherence and the same outcomes. Mixed methods process evaluation will be conducted. Post-training and post-follow-up qualitative focus group interviews will be conducted; facilitators, barriers, and mediators will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents,
2. ethnic Chinese aged 18-65 years with the ability to communicate in Cantonese or Putonghua,
3. who fulfil the DSM-5 diagnostic criteria for insomnia disorder according to a validated diagnostic tool, the Brief Insomnia Questionnaire (we include primary insomnia because it is more homogenous and less complicated than comorbid insomnia; if ZTEx is found to be effective for primary insomnia, then comorbid insomnia can be targeted in future studies),
4. scored at least 10 points in the Insomnia Severity Index,
5. are ambulant and can independently perform daily activities,
6. are physically inactive, defined as not having participated in at least 150 min of moderate intensity or 75 min of vigorous intensity physical activity a week, or the equivalent combination over the previous 3 months by self-report
7. have a smartphone compatible with WhatsApp, and
8. willing to give informed consent

Exclusion Criteria:

1. any current diagnosis fulfilling the DSM-IV criteria of a major depressive disorder, generalized anxiety disorders, post-traumatic stress disorder, panic disorder, substance use disorders, or schizophrenia as screened using the Chinese version of the Structured Clinical Interview for DSM-IV;
2. other sleep disorders, including circadian rhythm disorder, narcolepsy, obstructive sleep apnoea (OSA), and restless leg syndrome (RLS)/periodic leg movement disorder (PLMD) as determined based on cut-off scores (≥ 7 on narcolepsy; ≥ 8 on circadian rhythm disorder; ≥ 15 on OSA; ≥ 7 on RLS/PLMD) using SLEEP-50. If in doubt, subjects will be referred to our team psychiatrist (KF Chung) for further assessment;
3. any current medical conditions or side-effects of medication that are contributing significantly to the subject's insomnia;
4. taking medications or currently participating in other psychotherapies for insomnia or other psychiatric disorders;
5. impaired cognitive functioning (<22 points in HK-MoCA) or with difficulty in giving consent or understanding instructions;
6. pregnant;
7. shift work;
8. whose physical condition is such that physicians recommend that they refrain from exercising; and
9. fulfilling the criterion for obesity for Asians (body mass index, of 27.5 or above)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in the Insomnia Severity Index score | Baseline, week 8, week 16, week 24
  The subjects rate the severity of insomnia, the distress, and the functional impairment associated with insomnia on a 5-point scale. The score ranges from 0 to 28. The higher the score, the worse the outcome is.

SECONDARY OUTCOMES:
Sleep diary (7-day) | baseline, week 8, week 16, week 24
  The standardized sleep diary records the daily bedtime and rising time, from which the total time in bed (TIB) can be calculated.
Hospital Anxiety and Depression Scale | baseline, week 8, week 16, week 24
  The Hospital Anxiety and Depression Scale is a 14-items self-administered questionnaire, which assesses the severity of depressive and anxiety symptoms. The score ranges between 0 and 21 for either anxiety or depression. The higher the score, the worse the outcome is.
Multidimensional fatigue inventory-20 | baseline, week 8, week 16, week 24
  Multidimensional fatigue inventory-20 is a 20-items self-report instrument designed to measure severity of fatigue. The score ranges from 20 to 100. The higher the score, the worse the outcome is.
Actigraphy (7-day) | baseline, week 8, week 16, week 24
  Actigraphy measures wrist movements to assess sleep or waking state, is accomplished through an accelerometer in a wrist worn device.
Accelerometer (7-day) | baseline, week 8, week 16, week 24
  Accelerometer measures wrist movements to assess the physical activity levels.
Change in WAIS-IV Color Trails Test | baseline, week 8, week 16, week 24
  Change in Wechsler Adult Intelligence Scale, 4th edition (WAIS-IV) Color Trails Test score will be used to measure the attention function.
Change in WAIS-IV Stroop color-word Test | baseline, week 8, week 16, week 24
  Change in Wechsler Adult Intelligence Scale, 4th edition (WAIS-IV) Stroop color-word Test score will be used to measure the attention function.
Change in Digit Span-backward test | baseline, week 8, week 16, week 24
  Change in Digit Span-backward and forward test score will be used to measure the memory function.
Change in the Wisconsin Card Sorting Test | baseline, week 8, week 16, week 24
  Change in the Wisconsin Card Sorting Test score will be used to measure the executive function

OTHER OUTCOMES:
Intervention adherence (7 day) | week 1-8, week 12-15, week 20-23
  Patients will be told to record their daily physical activities or sleep health hygiene compliance onto the log.

CONTACTS AND LOCATIONS:
Overall Officials: WF Yeung, Principal Investigator — School of Nursing, the Hong Kong Polytechnic University
Locations (1):
- School of Nursing, the Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeung WF, Lai AY, Yu BY, Ho FY, Chung KF, Ho JY, Suen LK, Ho LM, Lam TH. Effect of zero-time exercise on physically inactive adults with insomnia disorder: A randomized controlled trial. Int J Nurs Stud. 2025 May;165:105033. doi: 10.1016/j.ijnurstu.2025.105033. Epub 2025 Feb 18. PMID 39999728